CLINICAL TRIAL: NCT05156073
Title: Shared Decision Making About Medication Use for People With Multiple Health Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Reading Hospital Family Health Care Center (Unknown); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00253480; K23AG054742 (NIH)
Record Dates: First submitted 2021-12-01; First posted 2021-12-14 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Polypharmacy; Dementia; Multiple Chronic Conditions; Deprescribing; Mild Cognitive Impairment
Keywords: Deprescribing; Dementia
MeSH Terms: conditions — Dementia; Multiple Chronic Conditions; Cognitive Dysfunction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The intervention consists of providing educational materials on deprescribing to:
  1. Patient and care partner cohort
  2. Primary care physician cohort
  Interventions: Other: Educational Materials

INTERVENTIONS:
Other: Educational Materials — 1. Patient care partner cohort:
     a. mailing of an educational brochure introducing deprescribing to patients with mild cognitive impairment or dementia and/or MCC and MCC care partners.
  2. Primary care physician cohort:
     1. education on deprescribing through a 15-45-minute presentation
     2. one-page weekly tip sheets on options for deprescribing in specific clinical situations and suggested language for deprescribing conversations.

SUMMARY:
The Shared Decision Making about Medication Use for People with Multiple Health Problems study will assess the feasibility and acceptability of a deprescribing educational intervention in primary care for patients with mild cognitive impairment or dementia and/or multiple chronic conditions (MCC), the patients' care partners, clinicians, and medical assistants.

The intervention consists of the following strategies: 1) a patient/caregiver component focused on education and activation about deprescribing, and 2) a clinician component focused on increasing clinician awareness about options and processes for deprescribing in the MCI/dementia and/or MCC population. Clinicians will each be asked to participate in a single, 15-minute educational session on deprescribing, and medical residents will receive a 45-minute lecture. Patients, caregivers, clinicians, and medical assistants will participate in a single one-on-one debriefing interview.

DETAILED DESCRIPTION:
People living with dementia are prescribed more medications and have more complex medication regimens than people without dementia. These problems are exacerbated in people with dementia and multiple chronic conditions (MCC). Having multiple diseases simultaneously (e.g., diabetes and hypertension, and dementia) leads to the use of multiple drugs (polypharmacy) and potentially inappropriate medications, in which the risks of medications outweigh the benefits, or medications do not align with the patient's treatment goals. For individuals with dementia and MCC, taking more medications is associated with a greater risk of adverse drug events, drug interactions, and treatment burden. Medication regimen complexity is a major source of burden for family caregivers of people living with dementia and has been associated with numerous adverse outcomes. Studies suggest that as many as 56% of people with dementia take at least one potentially inappropriate medication, including medications that can negatively affect cognitive function. Optimizing medication use through deprescribing (the process of reducing or stopping the use of potentially inappropriate medications or medications unlikely to be beneficial) can improve outcomes for patients with dementia and MCC. Therefore, the investigator proposes a patient-centered deprescribing educational intervention for older adults with mild cognitive impairment or dementia and/or MCC, generalizable to a range of primary care settings. This study builds on OPTIMIZE, a multisite randomized trial within Kaiser Permanente Colorado that has been recently completed. OPTIMIZE is the investigator team's primary care-based deprescribing intervention for patients with mild cognitive impairment and dementia, and MCC. OPTIMIZE consists of a patient and family component focused on education and activation about deprescribing and a clinician component to increase awareness about processes and language for deprescribing.

The investigators propose a pilot study of medication optimization through increased awareness of deprescribing for older adults with cognitive impairment and/or MCC. The intervention will have two components: a patient/ care partner component focused on education and activation about deprescribing, and a clinician component focused on increasing clinician awareness about options and processes for deprescribing in the cognitive impairment-MCC population. The proposed intervention has the following aims:

1. To establish the feasibility and acceptability of the intervention among patients, caregivers, clinicians, and medical assistants in one healthcare system by assessing:

   a. Acceptability and process measures from a qualitative analysis of debriefing interviews with patients, care partners, clinicians, and medical assistants.
2. To determine the preliminary efficacy of the intervention by assessing:

   1. Clinical documentation of deprescribing, defined as medication discontinuation or dose reduction.
   2. Clinical documentation of a discussion about medication appropriateness, safety, or effectiveness (yes/possible vs. no/absent).

ELIGIBILITY:
Inclusion Criteria:

This study has two cohorts: A Mild Cognitive Impairment (MCI)/Dementia cohort and a non-dementia cohort.

MCI/Dementia cohort:

* Age 65 or greater
* Diagnosis of MCI or dementia from International Classification of Diseases ICD-9 and ICD-10 codes
* At least one other chronic condition
* Five or more chronic medications (to include all prescription and over-the-counter medications, both scheduled and as needed)
* Have a primary care physician at the pilot clinic who has enrolled in the study
* Have a routine, scheduled visit with a primary care physician during the pilot study period (not an urgent, acute or pre-op visit)
* Patient must be able to hear well enough to participate in interviews on the telephone.

Non-dementia cohort:

* Age 75 or older
* No MCI or dementia diagnosis
* At least two chronic conditions documented
* 5 or more chronic medications (to include all prescription and over-the-counter medications, both scheduled and as needed)
* Have a primary care physician at the pilot clinic who has enrolled in the study
* Have a routine, scheduled visit with a primary care physician during the pilot study period (not an urgent, acute, or pre-op visit).
* Patient must be able to hear well enough to participate in interviews on the telephone.

Care partners:

* Age 21 years or greater
* Must be able to hear well enough to participate in interviews on the telephone.

Primary care physicians and medical assistants:

• All primary care physicians and medical assistants at the pilot site will be included. Physicians who only provide urgent care will be excluded.

Exclusion Criteria:

* As the pilot will be based in primary care, individuals residing in long-term care facilities or enrolled in hospice care at baseline will be excluded.
* Patients taking 4 or fewer different medications for all their health needs will be excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Green, MD, MPH, PhD, Principal Investigator — Johs Hopkins University
Locations (1):
- Reading Hospital Family Health Care Center, Reading, Pennsylvania, United States

REFERENCES:
- [Background] Boyd CM, Darer J, Boult C, Fried LP, Boult L, Wu AW. Clinical practice guidelines and quality of care for older patients with multiple comorbid diseases: implications for pay for performance. JAMA. 2005 Aug 10;294(6):716-24. doi: 10.1001/jama.294.6.716. PMID 16091574
- [Background] Alzheimer's Association. 2016 Alzheimer's disease facts and figures. Alzheimers Dement. 2016 Apr;12(4):459-509. doi: 10.1016/j.jalz.2016.03.001. PMID 27570871
- [Background] Lin PJ, Fillit HM, Cohen JT, Neumann PJ. Potentially avoidable hospitalizations among Medicare beneficiaries with Alzheimer's disease and related disorders. Alzheimers Dement. 2013 Jan;9(1):30-8. doi: 10.1016/j.jalz.2012.11.002. PMID 23305822
- [Background] Kelley AS, McGarry K, Gorges R, Skinner JS. The burden of health care costs for patients with dementia in the last 5 years of life. Ann Intern Med. 2015 Nov 17;163(10):729-36. doi: 10.7326/M15-0381. Epub 2015 Oct 27. PMID 26502320
- [Background] Willson MN, Greer CL, Weeks DL. Medication regimen complexity and hospital readmission for an adverse drug event. Ann Pharmacother. 2014 Jan;48(1):26-32. doi: 10.1177/1060028013510898. Epub 2013 Nov 5. PMID 24259639
- [Background] Bayliss EA, Shetterly SM, Drace ML, Norton J, Green AR, Reeve E, Weffald LA, Wright L, Maciejewski ML, Sheehan OC, Wolff JL, Gleason KS, Kraus C, Maiyani M, Du Vall M, Boyd CM. The OPTIMIZE patient- and family-centered, primary care-based deprescribing intervention for older adults with dementia or mild cognitive impairment and multiple chronic conditions: study protocol for a pragmatic cluster randomized controlled trial. Trials. 2020 Jun 18;21(1):542. doi: 10.1186/s13063-020-04482-0. PMID 32552857
- [Background] George J, Phun YT, Bailey MJ, Kong DC, Stewart K. Development and validation of the medication regimen complexity index. Ann Pharmacother. 2004 Sep;38(9):1369-76. doi: 10.1345/aph.1D479. Epub 2004 Jul 20. PMID 15266038
- [Background] Travis SS, Bernard MA, McAuley WJ, Thornton M, Kole T. Development of the family caregiver medication administration hassles scale. Gerontologist. 2003 Jun;43(3):360-8. doi: 10.1093/geront/43.3.360. PMID 12810899

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention (Deprescribing Education): The intervention consists of providing educational materials on deprescribing to:
  1. Patient and care partners, including the mailing of an educational brochure introducing deprescribing to patients with mild cognitive impairment or dementia and/or MCC and MCC care partners.
  2. Primary care physicians, including education on deprescribing through a 15-45-minute presentation and one-page weekly tip sheets on options for deprescribing in specific clinical situations and suggested language for deprescribing conversations.
Period: Overall Study
Arm/Group | Intervention (Deprescribing Education)
Started | 22
Completed | 21
Not Completed | 1
Not completed — Patient canceled appointment with PCP | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intervention (Deprescribing Education)
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.5 (7.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 8
Medications Prescribed to the Patient [Mean (Standard Deviation); unit: medications] | 13.3 (5.46)

OUTCOME MEASURES:

1. Primary Outcome: Preliminary Efficacy of the Intervention to be Assessed From Primary Care Clinician's Intervention Visit Clinical Notes and EHR
Description: The investigators will assess the impact of the intervention by assessing the primary care clinician's documentation from the clinic visit immediately after the patient and care partner receive the intervention brochure.
  The following will be evaluated:
  1. Primary care clinician's documentation of discussions about medication appropriateness, safety, or effectiveness.
  2. Primary care clinician's documentation of planned medication changes (new medications to be added, dose increases, dose reductions, or medications to be stopped).
  3. The proportion of patients who deprescribe one or more medications
  4. The proportion of patients who add one or more medications
  These measures will be extracted from the electronic medical record.
Time Frame: 1 year
Population: A total of 22 participants were enrolled and received the intervention brochure by mail. Data on clinical documentation was not available for two participants, therefore a total of 20 participants were analyzed in rows 1-4. Additionally, medication data was missing for three more participants in rows 5-6, thus a total of 17 participants were included in the analysis of rows 5-6.
Measure: Count of Participants; unit: Participants
Groups:
- Intervention (Deprescribing Education): The intervention consists of providing educational materials on deprescribing to:
  1. Patient care partner cohort, including the mailing of an educational brochure introducing deprescribing to patients with mild cognitive impairment or dementia and/or MCC and MCC care partners.
  2. Primary care physician cohort, including the education on deprescribing through a 15-45-minute presentation and one-page weekly tip sheets on options for deprescribing in specific clinical situations and suggested language for deprescribing conversations.
Arm/Group | Intervention (Deprescribing Education)
Number analyzed (Participants) | 20
Participants
  Documentation of a discussion about medication appropriateness, safety, or effectiveness | 15
  Documentation of any medications being discontinued | 7
  Documentation of a new medicine being started | 7
  Documentation of actions taken as part of the deprescribing process (e.g., order a blood test) | 7
  Proportion of patients who deprescribed 1+ medicines: number analyzed (Participants) | 17
  Proportion of patients who deprescribed 1+ medicines | 10
  The proportion of patients who added 1+ new medicine: number analyzed (Participants) | 17
  The proportion of patients who added 1+ new medicine | 10

2. Secondary Outcome: Acceptability of the Intervention to be Assessed Qualitatively From Debriefing Interviews
Description: The investigators will evaluate the acceptability of the intervention among patients, care partners, clinicians, and medical assistants by:
  a) determining which materials and features of the intervention are most and least acceptable to clinicians, medical assistants, patients, and care partners.
  These data will be obtained through the qualitative analysis of debriefing interviews.
Time Frame: 1 year
Population: Data Not Collected
Arm/Group | Intervention (Deprescribing Education)
Number analyzed (Participants) | 0

3. Secondary Outcome: Feasibility of the Intervention to be Assessed Qualitatively From Debriefing Interviews
Description: The investigators will evaluate the feasibility of the intervention among patients, care partners, clinicians, and medical assistants by:
  a) identifying features of the clinic's culture or workflow that served as barriers or facilitators of the intervention.
  These data will be obtained through the qualitative analysis of debriefing interviews.
Time Frame: 1 year
Population: Data Not Collected
Arm/Group | Intervention (Deprescribing Education)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 60 days
Groups:
- Intervention (Deprescribing Education): The intervention consists of providing educational materials on deprescribing to:
  1. Patient care partner cohort, including mailing of an educational brochure introducing deprescribing to patients with mild cognitive impairment or dementia and/or MCC and MCC care partners.
  2. Primary care physician cohort, including education on deprescribing through a 15-45-minute presentation and one-page weekly tip sheets on options for deprescribing in specific clinical situations and suggested language for deprescribing conversations.
Arm/Group | Intervention (Deprescribing Education)
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 3/22
Other Adverse Events (participants affected / at risk) | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (Deprescribing Education) (N=22)
Hospitalization (General disorders) | 2 (3)
Emergency Department Visit (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT05156073/Prot_000.pdf